CLINICAL TRIAL: NCT04139720
Title: Development and Effectiveness Verification of Sexual Harassment Prevention Via Education E-Book for Nursing: Randomized Controlled Experiments
Brief Title: Sexual Harassment Prevention for Nursing Via E-Book
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ya-Ling Tzeng, Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMUH108-REC1-086
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Sexual Harassment
Keywords: sexual harassment prevention; nurse; education; e-book
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Intervention Model Description: The repeated measurements randomization control trial will be used for the experimental design. We design a 45-minute course and 15 minutes of Q&A. Based on the gender in recruitment, the study used block randomization, and randomly assign participants who meet the selection criteria to the experimental group and the control group (1:1 ratio) by Random Allocation Software random assignment table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-book (Experimental): e-book learning mode of sexual harassment prevention training
  Interventions: Behavioral: e-book
- audio-visual and booklet (No Intervention): sexual harassment prevention audio-visual and booklet learning mode

INTERVENTIONS:
Behavioral: e-book — sexual harassment prevention via education e-book
  Arms: e-book

SUMMARY:
Nursing staff work closely with people and often have direct physical contact with patients, hence, they are high-risk individuals of sexual harassment. In particular for inexperienced newly employed nurses, if sexual harassment happened and without appropriate management, it may negatively impact physical and mental health, and even affect their willingness to engage in nursing field in the future. Therefore, how to assist the newly employed nurses to have the knowledge and ability to deal with sexual harassment in the workplace is important. Based on this, this study aims to improve the knowledge and practical ability of sexual harassment prevention, and develop "newly employed nurses' sexual harassment prevention training e-book" to implement gender perspective into nursing education which is in line with nursing clinical practice. The experimental research design is randomized controlled repeated measures; compare the differences between the two groups before and after the study to verify the effectiveness of the intervention. Overall, if it is proved effective, which will be able to enhance newly employed nurses' awareness of clinical sexual harassment and the ability to handle related incidents. The development of sexual harassment prevention materials can become a learning aid for nursing education. In addition to helping to reduce the adverse effects of sexual harassment in the nursing workplace, it will also help to establish the attention and consensus of the nursing profession on sexual harassment prevention.

DETAILED DESCRIPTION:
1. Research design: The repeated measurements randomization control trial is used for the study design. We design a 45-minute course and 15 minutes Q&A to enable learners to integrate knowledge and experience to achieve meaningful and valuable learning experiences by exploring problems, summarizing and integrating information and expression. After the end of the study, quantitative analysis was used to compare the differences between the experimental group and the control group before and after the study and two weeks later to verify the effectiveness of different learning models. In order to avoid the difference between the retest effect and the practice effect, the second post-test will be performed two weeks after the pre-test to balance the bias caused by the test tool. They used different learning models. The experimental group used the e-book learning mode of sexual harassment prevention training, the control group used the sexual harassment prevention audio-visual learning mode, the dependent variable is the sexual harassment prevention knowledge, and the sexual harassment event coping skill, sexual harassment incident management and sexual harassment learning motivation.
2. Randomization Process: The study used block randomization, and randomly assign participants who meet the selection criteria to the experimental group and the control group (1:1 ratio) by Random Allocation Software random assignment table. In addition, using the electronic form system, participants fill in the study number to replace the identifiable name, and then the research assistant uses the random distribution software to obtain a random assignment table, and use the table to allocate experimental and control group before the experiment. The sealed envelopes numbered 1 to 104 were arranged in the order of the groups. On the day of the study, the researchers take out the envelopes and assigned them to the participants according to the order of handing in the consents. Based on the group number (1 or 2) on the envelope bag, participants enter the designated meeting room for research.
3. Sample size calculation: This study uses the repeated measures of G-Power 3.1.9 windows and between factors among groups to calculate the sample size. According to the predecessor study, the power value is set to .8, the alpha value is set to .05, and the effect size (ES) value is .25 (moderate ES). The number of samples was 43 in the experimental group and 43 in the control group, a total of 86. If the loss rate was 20%, the total requirement participants are 104. According to the literature, male nursing staff accounted for around 3%, so 4 of them were male nurses.

sexual harassment coping skill

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20 years old
2. Nursing school graduation
3. full time job

Exclusion Criteria:

1. Not directly in contact with the patient, such as the supply room
2. Not engaged in nursing clinical work, such as research assistants

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
sexual harassment prevention knowledge | The experimental group and the control group will take the test after the intervention immediately.
  using Likert seven-point scale, scoring from 7 (totally agree) to 1 (totally disagree), the score range from 16-112 points, the higher the total score of the scale, the better the understanding of harassment prevention concept.
sexual harassment event coping skill | The experimental group and the control group will take the test after the intervention immediately.
  Includes: Enhancing personal processing coping strategies for sexual harassment (4 questions), strengthening personal awareness and monitoring systems (13 questions), and strengthening social organization and policy development (14 questions). The scoring method: 0 (totally disagree) to 4 (very agree).
sexual harassment incident management | The experimental group and the control group will take the test after the intervention immediately.
  The scale is divided into verbal and non-verbal parts, which are summarized into three categories, namely, problem-solving, emotion and evaluation part, which total 37 questions according to the different attributes of the corresponding behavior. A score of 0 means never to 4 part means to always do 4 points means it always is. A higher score indicates that the more often new nursing might we to react

SECONDARY OUTCOMES:
Include learning motivation of sexual harassment | The experimental group and the control group will take the test after the intervention immediately.
  Contains the learner's attention to the teaching material (12 questions), relevance (9 questions), confidence (9 questions), satisfaction (6 questions) and other learning motivation, a total of 36 questions, use Likert five-point scale, scoring method from 5 (very agreeable) to 1 (very disagree), the score range from 36-180 points, the higher the total score of the scale, the stronger the motivation of learning.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Tzeng, PhD, Principal Investigator — China Medical University, Taiwan

REFERENCES:
- [Derived] Chang TS, Tzeng YL, Teng YK, Chen CH. Effectiveness of an e-book in enhancing knowledge, coping behaviors and preventive strategies for sexual harassment prevention among new nurses: A randomized controlled study. Nurse Educ Pract. 2025 Jan;82:104198. doi: 10.1016/j.nepr.2024.104198. Epub 2024 Nov 22. PMID 39612767